CLINICAL TRIAL: NCT01767064
Title: Nudging Guideline-concordant Antibiotic Prescribing Using Public Commitments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jason Doctor, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: USCalifornia; RC4AG039115 (NIH)
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Acute Respiratory Infections (ARIs)
Keywords: ARIs, antibiotics, public commitment, quality improvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posted commitment letter (Experimental): The poster-sized (18x24 inches) commitment letter, written at the 8th grade reading-level and displayed in English and Spanish, emphasize clinician commitment to guidelines for appropriate antibiotic prescribing and explain why antibiotics are not appropriate in many cases. These letters, featuring clinician photographs and signatures, are displayed in clinician exam rooms for a 16-week period.
  Interventions: Other: Posted commitment letter
- Control (No Intervention): Usual care with no posted letters.

INTERVENTIONS:
Other: Posted commitment letter
  Arms: Posted commitment letter

SUMMARY:
Inappropriate antibiotic prescribing for acute respiratory infections (ARIs) persists despite decades of intervention efforts. Negative outcomes of inappropriate antibiotics include increased costs of care, adverse drug reactions, and rising prevalence of antibiotic-resistant bacteria. To address this public health problem, we apply the principles of commitment and consistency in an effort to influence clinician decision-making through the implementation of a low-cost behavioral "nudge" in the form of a simple public commitment device. Clinicians were asked to post in their exam room a signed letter indicating their commitments to reducing inappropriate antibiotic use for ARIs. Our hypothesis is that clinicians displaying the poster-sized commitment letters will decrease their inappropriate antibiotic prescribing for ARIs as compared to clinicians in the control condition (with no posted letter).

ELIGIBILITY:
Inclusion Criteria:

* Medical professionals licensed to provide care and prescribe medications (including antibiotics)
* Treating adult patients (18 years of age and older) from 5 Los Angeles community clinics

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason N Doctor, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- QueensCare Family Clinics, Los Angeles, California, United States

REFERENCES:
- [Derived] Meeker D, Knight TK, Friedberg MW, Linder JA, Goldstein NJ, Fox CR, Rothfeld A, Diaz G, Doctor JN. Nudging guideline-concordant antibiotic prescribing: a randomized clinical trial. JAMA Intern Med. 2014 Mar;174(3):425-31. doi: 10.1001/jamainternmed.2013.14191. PMID 24474434

RESULTS

PARTICIPANT FLOW:
Groups:
- Posted Commitment Letter: The poster-sized (18x24 inches) commitment letter, written at the 8th grade reading-level and displayed in English and Spanish, emphasize clinician commitment to guidelines for appropriate antibiotic prescribing and explain why antibiotics are not appropriate in many cases. These letters, featuring clinician photographs and signatures, are displayed in clinician exam rooms for a 16-week period.
  Posted commitment letter
Period: Overall Study
Arm/Group | Posted Commitment Letter | Control
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Clinicians
Groups:
- Total: Total of all reporting groups
Arm/Group | Posted Commitment Letter | Control | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (12.9) | 55 (9.5) | 54.3 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Inappropriate Antibiotic Prescribing for Patients With Acute Respiratory Infections (ARI)
Description: Using data from electronic health records, we will calculate clinician antibiotic prescribing rates for antibiotic-inappropriate ARI diagnoses: acute nasopharyngitis (ICD-9 460.x), acute laryngitis without obstruction (465.8), acute laryngopharyngitis (465.0), acute bronchitis (466.x), acute upper respiratory infections of other multiple sites (465.8), acute upper respiratory infections not otherwise specified (465.9), bronchitis not specified as acute or chronic (490.x), non-streptococcal pharyngitis (462.xx), and influenza with other respiratory manifestations (487.1). To control for temporal trends in antibiotic prescribing and provider-fixed effects, we will fit a logistic mixed effects model that predicts inappropriate antibiotic prescribing as a function of study arm and an indicator for baseline versus intervention period (a difference-in-differences regression).
Time Frame: up to 12 months post intervention
Population: clinicians
Measure: Number (95% Confidence Interval); unit: inappropriate prescribing events
Arm/Group | Posted Commitment Letter | Control
Number analyzed (Participants) | 7 | 7
inappropriate prescribing events | 33.7 [25.1 to 43.1] | 52.7 [44.2 to 61.9]

ADVERSE EVENTS:
Arm/Group | Posted Commitment Letter | Control
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes